CLINICAL TRIAL: NCT01997736
Title: A Pilot Study Evaluating the Safety and Effectiveness of the Toray Satake Balloon Thermal Ablation System for the Treatment of Paroxysmal Atrial Fibrillation
Brief Title: Pilot Study Evaluating the Toray Satake Balloon Thermal Ablation System for Treatment of Paroxysmal Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toray Industries (America), Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Toray America 2013-001
Record Dates: First submitted 2013-11-08; First posted 2013-11-28 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2018-04

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Paroxysmal Atrial Fibrillation; Catheter Ablation; Ablation Techniques
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Ablation (Experimental)
  Interventions: Device: Ablation

INTERVENTIONS:
Device: Ablation
  Other Names: Toray Satake Balloon Thermal Ablation System

SUMMARY:
The purpose of this study is to collect preliminary safety and effectiveness data evaluating the Toray Satake Balloon Thermal Ablation System (TSB)to treat subjects with symptomatic paroxysmal atrial fibrillation that is resistant to antiarrhythmic drug therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of recurrent symptomatic paroxysmal atrial fibrillation
* ≥2 Symptomatic atrial fibrillation episodes
* At least 1 paroxysmal atrial fibrillation episode documented by an ECG or device recording system in the 6 months prior to enrollment AND
* At least 1 additional (for a total of ≥2) paroxysmal atrial fibrillation episode documented by an ECG or device recording system, OR, at a minimum, a physician's note indicating recurrent symptomatic atrial fibrillation
* No episode >7 days
* Failed to respond to or is intolerant of ≥1 Class I, II, III or IV antiarrhythmic drug
* Able and willing to provide informed consent and Health Insurance Privacy and Portability Act (HIPAA) authorization
* Able and willing to meet all study requirements, including attending all post-ablation procedure assessments and visits

Exclusion Criteria:

* Left atrium ≥50 mm
* Chronically used amiodarone in the 3 months prior to enrollment
* Previous left atrial ablation or surgical treatment for atrial fibrillation
* Left ventricular ejection fraction (LVEF) <35 %
* New York Heart Association (NYHA) Class III or IV heart failure
* History of myocardial infarction (MI) or unstable angina in the 6 months prior to enrollment
* Multiple other exclusion criteria to establish overall good health and likely study compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-11-22 (Actual); Primary Completion 2015-09-15 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of major complications | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David Haines, MD, Principal Investigator — Corewell Health East
Locations (4):
- United States (4):
  - William Beaumont Hospital, Royal Oak, Royal Oak, Michigan
  - Mount Sinai Hospital, New York, New York
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Satake S, Tanaka K, Saito S, Tanaka S, Sohara H, Hiroe Y, Miyashita Y, Takahashi S, Murakami M, Watanabe Y. Usefulness of a new radiofrequency thermal balloon catheter for pulmonary vein isolation: a new device for treatment of atrial fibrillation. J Cardiovasc Electrophysiol. 2003 Jun;14(6):609-15. doi: 10.1046/j.1540-8167.2003.02577.x. PMID 12875422
- [Background] Sohara H, Satake S, Tanaka K, et al. Modification of electrophysiological properties of pulmonary veins and adjacent left atrial tissue by radiofrequency thermal balloon circumferential ablation around the pulmonary vein ostia: correlation with non-recurrence of atrial fibrillation. Journal of Arrhythmia 21(3):384-397, 2005.
- [Background] Sohara H, Takeda H, Ueno H, Oda T, Satake S. Feasibility of the radiofrequency hot balloon catheter for isolation of the posterior left atrium and pulmonary veins for the treatment of atrial fibrillation. Circ Arrhythm Electrophysiol. 2009 Jun;2(3):225-32. doi: 10.1161/CIRCEP.108.817205. Epub 2009 Apr 2. PMID 19808472
- [Background] Sohara H, Satake S, Takeda H, et al. Radiofrequency hot balloon catheter ablation for the treatment of atrial fibrillation: a 3-center study in Japan. Journal of Arrhythmia 29:20-27, 2013